CLINICAL TRIAL: NCT00883909
Title: ARI103094-Follow-Up Study for REDUCE Study Subjects
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 103094
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Neoplasms, Prostate
Keywords: Prostate Cancer; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PART B: Collection of tissue blocks or unstained slides from positive biopsies.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- observational: A follow-up study in adult male subjects who have received investigational
  Interventions: Drug: dutasteride

INTERVENTIONS:
Drug: dutasteride — A follow-up study in adult male subjects who have received investigational product

SUMMARY:
ARI103094 is a follow-up study in adult male subjects who have received investigational product (either dutasteride or placebo) in the REDUCE Study (REduction by DUasteride of prostate Cancer Events), ARI40006, A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of the Efficacy and Safety of Dutasteride 0.5mg Administered Orally Once Daily for Four Years to Reduce the Risk of Biopsy-Detectable Prostate Cancer. There are 2 parts to this REDUCE Follow-Up Study, Part A and Part B:

* REDUCE Follow-Up Study, Part A, is a 2 year observational study which will follow eligible subjects for 2 years after completion of the 4 Contact in the REDUCE study. Eligible subjects for Part A, the 2 Year Observational Study fall into 3 groups as follows: (1) REDUCE subjects who completed treatment with investigational product (dutasteride or placebo) through the REDUCE 4 Year study visit [Visit 10], (2) REDUCE subjects who developed prostate cancer, were withdrawn from investigational product and participated in Prostate Cancer follow-up until the REDUCE 4 Year study visit [Visit 10P] or (3) REDUCE subjects who were withdrawn from investigational product and participated in observational phone follow up until the REDUCE 4 Year phone call after withdrawing from IP (expected Visit 10). The objective of this observational study for eligible REDUCE subjects is to collect and summarize data on prostate cancer (the incidence of newly diagnosed prostate cancers and changes in prostate cancer diagnosed during the REDUCE study) and serious adverse events (SAEs) for 2 years beyond the prospectively planned 4 year double blind, placebo-controlled study, REDUCE.
* REDUCE Follow-Up Study, Part B, is for collection of cancer positive prostate biopsy tissue blocks/slides from subjects who were diagnosed with prostate cancer in the REDUCE study.

ELIGIBILITY:
Inclusion Criteria: PART A

* Any subject who has participated in the REDUCE Study and meets one of the following eligibility criteria is eligible for Part A, 2 Year Observational Follow-Up Study:
* Completed 4 years on Investigational Product through the REDUCE 4 Year study visit (Visit 10) OR
* Was diagnosed with prostate cancer during the REDUCE study, discontinued Investigational Product (IP) but participated in REDUCE Prostate Cancer Follow-Up visits through the 4 Year study visit (Visit 10P) OR
* Withdrew from REDUCE study visit participation and IP (for any reasons) but participated in REDUCE Follow-Up phone calls every 6 months through the 4 Year phone call

Exclusion Criteria: PART A Subjects meeting the following criterion must not be enrolled in Part A of the study

* Inability/unwillingness to participate in the Follow-Up Study phone calls.

Inclusion Criteria: PART B

Subjects eligible for enrolment in Part B of the study must meet the following criteria:

* Any subject who was diagnosed with prostate cancer based on a prostate biopsy during participation in the REDUCE Study, regardless of when their REDUCE study participation ended.

Exclusion Criteria: PART B

* The exclusion criterion only applies to Part A, the 2 year Observational Follow-Up Study. There are no exclusion criteria for Part B, Prostate Biopsy Tissue Study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without prostate cancer that participated in the REDUCE trial
Sampling Method: Probability Sample
Enrollment: 2795 (Actual)
Dates: Start 2009-04-09; Primary Completion 2010-12-01 (Actual); Study Completion 2010-12-29 (Actual)

PRIMARY OUTCOMES:
To collect and summarize data for 2 years beyond the prospectively planned 4 year double blind, placebo-controlled REDUCE study. | 2 years

SECONDARY OUTCOMES:
To collect and summarize data on Adverse Events for 2 years beyond the prospectively planned 4 year double blind, placebo-controlled REDUCE study. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (239):
- United States (71):
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Laguna Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, San Bernardino, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pinecrest, Florida
  - GSK Investigational Site, Pinellas Park, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Galesburg, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Greenwood, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Watertown, Massachusetts
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Sartell, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, West Orange, New Jersey
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Garden City, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Staten Island, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Sheffield, Ohio
  - GSK Investigational Site, Ponca City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Bala-Cynwyd, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, State College, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Myrtle Beach, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (3):
  - GSK Investigational Site, Av Córdoba 2424, Buenos Aires
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
- Canada (16):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Waterloo, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Granby, Quebec
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Finland (5):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Lappeenranta
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
- France (22):
  - GSK Investigational Site, Auch
  - GSK Investigational Site, Bourgoin
  - GSK Investigational Site, Cannes
  - GSK Investigational Site, Carpentras
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Longjumeau
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Mantes-la-Jolie
  - GSK Investigational Site, Montauban
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Orléans
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Ploemeur
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Martin-d'Hères
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Troyes
- Germany (53):
  - GSK Investigational Site, Backnang, Baden-Wurttemberg
  - GSK Investigational Site, Bruchsal, Baden-Wurttemberg
  - GSK Investigational Site, Neckargemünd, Baden-Wurttemberg
  - GSK Investigational Site, Aichach, Bavaria
  - GSK Investigational Site, Herzogenaurach, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Planegg, Bavaria
  - GSK Investigational Site, Tirschenreuth, Bavaria
  - GSK Investigational Site, Hagenow, Brandenburg
  - GSK Investigational Site, Hennigsdorf, Brandenburg
  - GSK Investigational Site, Oranienburg, Brandenburg
  - GSK Investigational Site, Senftenberg, Brandenburg
  - GSK Investigational Site, Strausberg, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hochheim am Main, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Seligenstadt, Hesse
  - GSK Investigational Site, Buchholz, Lower Saxony
  - GSK Investigational Site, Ganderkesee, Lower Saxony
  - GSK Investigational Site, Holzminden, Lower Saxony
  - GSK Investigational Site, Leer, Lower Saxony
  - GSK Investigational Site, Wismar, Mecklenburg-Vorpommern
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Erkrath, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Kempen, North Rhine-Westphalia
  - GSK Investigational Site, Langenfeld, North Rhine-Westphalia
  - GSK Investigational Site, Bad Bergzaben, Rhineland-Palatinate
  - GSK Investigational Site, Bad Schlema, Saxony
  - GSK Investigational Site, Bautzen, Saxony
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Döbeln, Saxony
  - GSK Investigational Site, Grimma, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Neustadt, Saxony
  - GSK Investigational Site, Plauen, Saxony
  - GSK Investigational Site, Radebeul, Saxony
  - GSK Investigational Site, Schwarzenberg, Saxony
  - GSK Investigational Site, Wilkau-Haßlau, Saxony
  - GSK Investigational Site, Zwickau, Saxony
  - GSK Investigational Site, Eisleben Lutherstadt, Saxony-Anhalt
  - GSK Investigational Site, Gardelegen, Saxony-Anhalt
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Hettstedt, Saxony-Anhalt
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lauenburg, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Plön, Schleswig-Holstein
  - GSK Investigational Site, Gotha, Thuringia
  - GSK Investigational Site, Ilmenau, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (6):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Periohi Dragana, Alexandroupolis
  - GSK Investigational Site, Rhodes
  - GSK Investigational Site, Thessaloniki
- Netherlands (12):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Arnhem
  - GSK Investigational Site, Capelle aan den IJssel
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Roermond
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Tilburg
- Spain (24):
  - GSK Investigational Site, Alava
  - GSK Investigational Site, Alcala de Henares (Madrid)
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Ciudad Real
  - GSK Investigational Site, Don Benito (Badajoz)
  - GSK Investigational Site, Galdakano
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Ibiza Town
  - GSK Investigational Site, La Laguna-Tenerife
  - GSK Investigational Site, Logroño
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Manacor (Palma de Mallorca)
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Sagunto
  - GSK Investigational Site, San Sebastián
  - GSK Investigational Site, Sant Joan d'Alacant
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Soria
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
- Sweden (11):
  - GSK Investigational Site, Borås
  - GSK Investigational Site, Eskilstuna
  - GSK Investigational Site, Gävle
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Karlshamn
  - GSK Investigational Site, Kristianstad
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Östersund
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Umeå
  - GSK Investigational Site, Vålberg
- United Kingdom (15):
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Exeter, Devon
  - GSK Investigational Site, Plymouth, Devon
  - GSK Investigational Site, Buckshaw Village, Chorley, Lancashire
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Chichester, Sussex West
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Clydebank, Glasgow
  - GSK Investigational Site, Edgbaston, Birmingham
  - GSK Investigational Site, High Heaton, Newcastle Upon Tyne
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, Torquay
  - GSK Investigational Site, Waterloo, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Grubb RL, Andriole GL, Somerville MC, Mahoney C, Manyak MJ, Castro R. The REDUCE Follow-Up Study: low rate of new prostate cancer diagnoses observed during a 2-year, observational, followup study of men who participated in the REDUCE trial. J Urol. 2013 Mar;189(3):871-7. doi: 10.1016/j.juro.2012.09.099. Epub 2012 Sep 25. PMID 23021996
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 103094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 103094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 103094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 103094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 103094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 103094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 103094 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register